CLINICAL TRIAL: NCT05626881
Title: Evaluation of the Efficacy and Tolerability of Autologous Intralesional Platelet-rich Plasma, Topical Silymarin, and Combined Autologous Intralesional Platelet-rich Plasma With Topical Silymarin in the Treatment of Melasma
Brief Title: Efficacy of Intralesional PRP +/- Topical Silymarin in the Treatment of Melasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Kamal Shaker, Resident physician at Dermatology department, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-04-08
Record Dates: First submitted 2022-10-17; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP group (Active Comparator): It will include patients with melasma treated with PRP sessions every two weeks for three monthsPRP is injected intralesionally at the site of melasma using a 30 G hypodermic needle through an insulin syringe. A maximum of 2.0 ml of PRP will be injected into the dermis (about 1.5-2.0 mm deep) about 1 cm apart to raise dermal papules
  Interventions: Drug: PRP
- Silymarin group (Active Comparator): It will include patients with melasma applying with topical Silymarin cream. Silymarin cream will be prepared in the Faculty of Pharmcy according to the following formulation: stearic acid 15 g, glycerin 5 g, KOH 0.72 g, H2O 79 g, sodium benzoate (0.1%), and Tween-80 (1%). Silymarin was manufactured with concentration of 1.4%. Silymarin will be applied twice daily. The duration of treatment will be 3 months.
  Interventions: Drug: sylimarin cream
- PRP + silymarin group (Active Comparator): It will be treated by using both PRP sessions and applying topical Silymarin cream. Silymarin will be applied twice daily, while PRP sessions every 2 weeks.
  Interventions: Drug: PRP; Drug: sylimarin cream

INTERVENTIONS:
Drug: PRP — It will include patients with melasma treated with PRP sessions every two weeks for three months. 10 ml of venous blood will withdraw by means of a wide bore needle and a vacutainer containing an anticoagulant (Acid citrate dextrose).
  Double centrifugation will be done. First centrifugation, will be done for 10 minutes. After the first centrifugation, three layers will be seen , Second centrifugation will be done for 10 min, after which the platelets separate and form a grayish pellet at the bottom of the tube and the rest will be platelet-poor plasma. About 1 ml of this platelet-poor plasma will be decanted off and the platelet pellet will be resuspended in the remaining plasma to get PRP. With 10 ml blood, about 1-1.5 ml of PRP will be obtained.
  PRP is injected intralesionally at the site of melasma using a 30 G hypodermic needle through an insulin syringe.
  Arms: PRP + silymarin group; PRP group
Drug: sylimarin cream — Silymarin was manufactured with concentration of 1.4%
  Arms: PRP + silymarin group; Silymarin group

SUMMARY:
Melasma is an acquired disorder of melanogenesis leading to hyperpigmentation and manifested by symmetrical brown to gray-black macules and patches with serrated irregular edges . It occurs especially in sun-exposed areas and affects young to middle-aged women. It is most commonly seen on the face and less commonly on the neck, arms, and chest . Platelet rich plasma (PRP) is defined as a small volume of autologous plasma that contains a high concentration of platelets obtained by centrifugation of autologous blood and subsequent suspension of platelets

ELIGIBILITY:
Inclusion Criteria:

* Females in the reproductive age (18 years old and above) presented with melasma confirmed by wood's light.

Exclusion Criteria:

* Pregnant and lactating.
* Systemic diseases that may cause facial hyperpigmentation (e.g: thyroid diseases, renal, hepatic or endocrinal disorders).
* Patients receiving depigmenting drugs oral or topical in previous 3 months, drugs that prolong bleeding as aspirin, hormone replacement therapy or contraceptive pills.
* Patients with anemia, thrombocytopenia, coagulopathies or patient on anticoagulant therapy and patients with iron deficiency.
* Patient with infections in the face e.g. herpes.
* Patients with history of scarring or keloid formation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in mMASI SCORE | 8 months
  The mMASI score is calculated by subjective assessment of 3 factors: area (A) of involvement, darkness (D), and homogeneity (H), with the forehead (f), right malar region (rm), left malar region (lm), and chin (c), corresponding to 30%, 30%, 30%, and 10% of the total face, respectively. The area of involvement in each of these 4 areas is given a numeric value of 0 to 6 (0 = no involvement; 1 = \10%; 2 = 10%-29%; 3 = 30%-49%; 4 = 50%-69%; 5 = 70%-89%; and 6 = 90%- 100%). Darkness and homogeneity are rated on a scale from 0 to 4 (0 = absent; 1 = slight; 2 = mild; 3 = marked; and 4 = maximum). The MASI score is calculated by adding the sum of the severity ratings for darkness and homogeneity, multiplied by the value of the area of involvement, for each of the 4 facial areas.
  The total score range is 0 to 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sarkar R, Arora P, Garg VK, Sonthalia S, Gokhale N. Melasma update. Indian Dermatol Online J. 2014 Oct;5(4):426-35. doi: 10.4103/2229-5178.142484. PMID 25396123
- [Background] Cestari TF, Dantas LP, Boza JC. Acquired hyperpigmentations. An Bras Dermatol. 2014 Jan-Feb;89(1):11-25. doi: 10.1590/abd1806-4841.20142353. PMID 24626644
- [Background] Achar A, Rathi SK. Melasma: a clinico-epidemiological study of 312 cases. Indian J Dermatol. 2011 Jul;56(4):380-2. doi: 10.4103/0019-5154.84722. PMID 21965843
- [Background] Sirithanabadeekul P, Dannarongchai A, Suwanchinda A. Platelet-rich plasma treatment for melasma: A pilot study. J Cosmet Dermatol. 2020 Jun;19(6):1321-1327. doi: 10.1111/jocd.13157. Epub 2019 Sep 30. PMID 31568636